CLINICAL TRIAL: NCT06148181
Title: A Randomized, Double-blind, Placebo-controlled, Phase 1a Study to Evaluate the Safety and Pharmacokinetics of Single Ascending Doses of ABBV-141 in Healthy Adult Western and Asian Subjects
Brief Title: A Study to Evaluate Adverse Events and How Single Ascending Doses of ABBV-141 Move Through the Body of Healthy Adult Western and Asian Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Basic Science
Other Study IDs: M24-693
Record Dates: First submitted 2023-11-20; First posted 2023-11-28 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: Healthy Volunteers
Keywords: ABBV-141; Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (8):
- Part 1, ABBV-141 (Intravenous [IV]) (Experimental): Western participants will receive a single IV dose of ABBV-141.
  Interventions: Drug: ABBV-141
- Part 1, Placebo for ABBV-141 (IV) (Placebo Comparator): Western participants will receive a single IV dose of placebo for ABBV-141.
  Interventions: Drug: Placebo for ABBV-141
- Part 1, ABBV-141 (subcutaneous [SC]) (Experimental): Western participants will receive a single SC dose of ABBV-141.
  Interventions: Drug: ABBV-141
- Part 1, Placebo for ABBV-141 (SC) (Placebo Comparator): Western participants will receive a single SC dose of placebo for ABBV-141.
  Interventions: Drug: Placebo for ABBV-141
- Part 2, ABBV-141 (IV) (Experimental): Asian participants will receive a single IV dose of ABBV-141.
  Interventions: Drug: ABBV-141
- Part 2, Placebo for ABBV-141 (IV) (Placebo Comparator): Asian participants will receive a single IV dose of placebo for ABBV-141.
  Interventions: Drug: Placebo for ABBV-141
- Part 2, ABBV-141 (SC) (Experimental): Asian participants will receive a single SC dose of ABBV-141.
  Interventions: Drug: ABBV-141
- Part 2, Placebo for ABBV-141 (SC) (Placebo Comparator): Asian participants will receive a single SC dose of placebo for ABBV-141.
  Interventions: Drug: Placebo for ABBV-141

INTERVENTIONS:
Drug: ABBV-141 — Infusion; intravenous (IV)
  Arms: Part 1, ABBV-141 (Intravenous [IV]); Part 2, ABBV-141 (IV)
Drug: Placebo for ABBV-141 — Infusion; IV
  Arms: Part 1, Placebo for ABBV-141 (IV); Part 2, Placebo for ABBV-141 (IV)
Drug: ABBV-141 — Injection; subcutaneous (SC)
  Arms: Part 1, ABBV-141 (subcutaneous [SC]); Part 2, ABBV-141 (SC)
Drug: Placebo for ABBV-141 — Injection; SC
  Arms: Part 1, Placebo for ABBV-141 (SC); Part 2, Placebo for ABBV-141 (SC)

SUMMARY:
The purpose of this study is to assess the safety, tolerability, pharmacokinetics (PK) and immunogenicity after single ascending doses (SAD) of ABBV-141 in healthy adult Western and Asian participants.

ELIGIBILITY:
Inclusion Criteria:

* A condition of general good health, based upon the results of a medical history, physical examination, vital signs, laboratory profile and a 12-lead electrocardiogram (ECG).
* Body Mass Index (BMI) is ≥ 18.0 to ≤ 32.0 kg/m2 after rounding to the tenths decimal.

For Part 2 only:

-Han Chinese ethnicity or Japanese ethnicity based on the following criteria:

* Han Chinese: First-generation Han Chinese with both parents of Han Chinese descent.
* Japanese: First- or second-generation Japanese with both parents and all four grandparents born in Japan and of Japanese descent.

Exclusion Criteria:

* History of epilepsy, any clinically significant cardiac, respiratory (except mild asthma as a child), renal, hepatic, gastrointestinal, hematologic, or psychiatric disease or disorder, or any uncontrolled medical illness.
* History of any clinically significant sensitivity or allergy to any medication, topical creams, or food.

Additionally for Part 1, only:

* Presence of foreign bodies, local irritation or infections, active skin diseases, tattoos, and/or scars on the thighs which may preclude the skin biopsy collection site planned as per schedule of activities.
* History of bruising easily, bleeding disorders, thrombocytopenia, or hypo-coagulation disorder.
* History of sensitivity to or allergies to adhesives or evidence of fragile or easily damaged skin.
* Evidence of hypertrophic scarring.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2024-01-29 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) of ABBV-141 | Up to Day 85
  Cmax of ABBV-141 will be assessed.
Time to Cmax (Tmax) of ABBV-141 | Up to Day 85
  Tmax of ABBV-141 will be assessed.
Area Under the Serum Concentration-time Curve (AUC) of ABBV-141 from time 0 to the time of last measurable concentration (AUCt) | Up to Day 85
  AUCt of ABBV-141 will be determined.
AUC of ABBV-141 from Time 0 to Infinity (AUCinf) | Up to Day 85
  AUCinf of ABBV-141 will be assessed.
Terminal Phase Elimination Rate Constant (β) of ABBV-141 | Up to Day 85
  Terminal phase elimination rate constant (β) of ABBV-141 will be assessed.
Terminal Phase Elimination Half-life (t1/2) of ABBV-141 | Up to Day 85
  Terminal phase elimination half-life (t1/2) of ABBV-141 will be assessed.
Dose Normalized Cmax of ABBV-141 | Up to Day 85
  Dose normalized Cmax of ABBV-141 will be assessed.
Dose Normalized AUC of ABBV-141 | Up to Day 85
  Dose normalized AUC of ABBV-141 will be assessed.
Number of Adverse Events (AEs) | Baseline to Day 85
  An adverse event (AE) is defined as any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product which does not necessarily have a causal relationship with this treatment.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (1):
- Acpru /Id# 261162, Grayslake, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=M24-693